CLINICAL TRIAL: NCT01513460
Title: A Multicenter, Randomized, Blinded, Active-controlled, Parallel-group Study to Compare the Efficacy, Tolerability and Safety of NVA237 Compared to Tiotropium Added on to Fluticasone/Salmeterol in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy, Tolerability and Safety of NVA237 in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNVA237AAU01
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease,; NVA 237,; glycopyrronium,; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- NVA237 + Fluticasone/Salmeterol (Flu/Sal) (Experimental): NVA237 50 µg once daily (NVA237 + Tiotropium placebo + Flu/Sal). NVA237 50 μg o.d., delivered via single-dose dry-powder inhaler (SDDPI) o.d. plus Placebo to tiotropium o.d. delivered via a proprietary inhalation device plus Flu/Sal 500/50 μg b.i.d. delivered via a proprietary inhalation device. In addition, at Visit 1, all participants were provided with a short acting β2-agonist (salbutamol) which they were instructed to use throughout the study as rescue medication.
  Interventions: Drug: NVA237 50µg once daily; Drug: Flu/Sal; Drug: NVA237 placebo + Tiotropium placebo.
- Tiotropium + Flu/Sal (Active Comparator): Tiotropium 18µg once daily (NVA237 placebo + Tiotropium + Flu/Sal). Tiotropium 18 μg o.d. delivered via a proprietary inhalation device plus Placebo to NVA237 o.d. delivered via single-dose dry-powder inhaler (SDDPI) plus Flu/Sal 500/50 μg b.i.d. delivered via a proprietary inhalation device. In addition, at Visit 1, all participants were provided with a short acting β2-agonist (salbutamol) which they were instructed to use throughout the study as rescue medication.
  Interventions: Drug: Tiotropium 18µg once daily; Drug: Flu/Sal; Drug: NVA237 placebo + Tiotropium placebo.
- Flu/Sal (Placebo Comparator): Placebo (NVA237 placebo + Tiotropium placebo + Flu/Sal). Placebo to tiotropium o.d. delivered via a proprietary inhalation device plus Placebo to NVA237 o.d. delivered via single-dose dry-powder inhaler (SDDPI) plus Flu/Sal 500/50 μg b.i.d. delivered via a proprietary inhalation device. In addition, at Visit 1, all participants were provided with a short acting β2-agonist (salbutamol) which they were instructed to use throughout the study as rescue medication.
  Interventions: Drug: Flu/Sal; Drug: NVA237 placebo + Tiotropium placebo.

INTERVENTIONS:
Drug: NVA237 50µg once daily — NVA237 50 μg o.d., delivered via single-dose dry-powder inhaler (SDDPI)
  Arms: NVA237 + Fluticasone/Salmeterol (Flu/Sal)
Drug: Tiotropium 18µg once daily — Tiotropium 18 μg o.d. delivered via a proprietary inhalation device
  Arms: Tiotropium + Flu/Sal
Drug: Flu/Sal — Flu/Sal 500/50 μg b.i.d. delivered via a proprietary inhalation device
Drug: NVA237 placebo + Tiotropium placebo. — Tiotropium 18 μg o.d. delivered via a proprietary inhalation device

SUMMARY:
This study will assess the efficacy, tolerability and safety of NVA237 compared to tiotropium when added on to fluticasone/salmeterol in patients with chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Moderate to Severe COPD (Stage II or Stage III) according to the GOLD 2010 guideline
* Current or ex-smokers who have a smoking history of at least 10 pack years
* Qualifying FEV1 at Visit 2 (day -7)

Exclusion Criteria:

* Patients with a history of asthma or a history of high blood eosinophil count (>600/mm³)
* Patients with concomitant pulmonary disease
* Patients with lung lobectomy or lung volume reduction or lung transplantation
* Patients with α-1 antitrypsin deficiency
* Patients who have had live attenuated vaccinations within 30 days prior to screening visit or during run-in period

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 773 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (67):
- Australia (56):
  - Novartis Investigative Site, Baulkham Hills, New South Wales
  - Novartis Investigative Site, Brookvale, New South Wales
  - Novartis Investigative Site, Castle Hill, New South Wales
  - Novartis Investigative Site, Dapto, New South Wales
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Ermington, New South Wales
  - Novartis Investigative Site, Gosford, New South Wales
  - Novartis Investigative Site, Hinchinbrook, New South Wales
  - Novartis Investigative Site, Kingswood, New South Wales
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Arundel, Queensland
  - Novartis Investigative Site, Aspley, Queensland
  - Novartis Investigative Site, Beenleigh, Queensland
  - Novartis Investigative Site, Browns Plains, Queensland
  - Novartis Investigative Site, Chemside, Queensland
  - Novartis Investigative Site, Deception Bay, Queensland
  - Novartis Investigative Site, Everton Plaza, Queensland
  - Novartis Investigative Site, Holland Park, Queensland
  - Novartis Investigative Site, Jimboomba, Queensland
  - Novartis Investigative Site, Kedron, Queensland
  - Novartis Investigative Site, Kenmore, Queensland
  - Novartis Investigative Site, Kippa-Ring, Queensland
  - Novartis Investigative Site, Logan Central, Queensland
  - Novartis Investigative Site, Loganholme, Queensland
  - Novartis Investigative Site, Mermaid Beach, Queensland
  - Novartis Investigative Site, Morayfield, Queensland
  - Novartis Investigative Site, Nerang, Queensland
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Daw Park, South Australia
  - Novartis Investigative Site, Glenelg East, South Australia
  - Novartis Investigative Site, Golden Grove, South Australia
  - Novartis Investigative Site, Hamley Bridge, South Australia
  - Novartis Investigative Site, Kensington Gardens, South Australia
  - Novartis Investigative Site, Prospect, South Australia
  - Novartis Investigative Site, Dandenong, Victoria
  - Novartis Investigative Site, Lalor, Victoria
  - Novartis Investigative Site, Malvern, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Noble Park, Victoria
  - Novartis Investigative Site, Oakleigh East, Victoria
  - Novartis Investigative Site, Preston, Victoria
  - Novartis Investigative Site, Rosebud, Victoria
  - Novartis Investigative Site, Bicton, Western Australia
  - Novartis Investigative Site, East Fremantle, Western Australia
  - Novartis Investigative Site, East Victoria Park, Western Australia
  - Novartis Investigative Site, Fremantle, Western Australia
  - Novartis Investigative Site, Mirrabooka, Western Australia
  - Novartis Investigative Site, Morley, Western Australia
  - Novartis Investigative Site, Nedlands, Western Australia
  - Novartis Investigative Site, Noranda, Western Australia
  - Novartis Investigative Site, Perth, Western Australia
  - Novartis Investigative Site, Pinjarra, Western Australia
  - Novartis Investigative Site, Spearwood, Western Australia
  - Novartis Investigative Site, Woodvale, Western Australia
  - Novartis Investigative Site, Yokine, Western Australia
- New Zealand (11):
  - Novartis Investigative Site, Auckland, New Zealand
  - Novartis Investigative Site, Christchurch, New Zealand
  - Novartis Investigative Site, Hamilton, New Zealand
  - Novartis Investigative Site, Tauranga, New Zealand
  - Novartis Investigative Site, Tauranga, Tauranga
  - Novartis Investigative Site, Wellington, Wellington Region
  - Novartis Investigative Site, Auckland
  - Novartis Investigative Site, Christchurch
  - Novartis Investigative Site, Dunedin
  - Novartis Investigative Site, Grafton, Auckland
  - Novartis Investigative Site, Wellington

REFERENCES:
- [Derived] Frith PA, Thompson PJ, Ratnavadivel R, Chang CL, Bremner P, Day P, Frenzel C, Kurstjens N; Glisten Study Group. Glycopyrronium once-daily significantly improves lung function and health status when combined with salmeterol/fluticasone in patients with COPD: the GLISTEN study, a randomised controlled trial. Thorax. 2015 Jun;70(6):519-27. doi: 10.1136/thoraxjnl-2014-206670. Epub 2015 Apr 3. PMID 25841237

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NVA237 + Fluticasone/Salmeterol (Flu/Sal) | Tiotropium + Flu/Sal | Flu/Sal
Started | 258 | 258 | 257
Full Analysis Set | 257 | 258 | 257
Per-protocol Set | 196 | 186 | 166
Completed | 229 | 226 | 201
Not Completed | 29 | 32 | 56
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Abnormal laboratory value | 1 | 0 | 1
Not completed — Lack of Efficacy | 1 | 2 | 5
Not completed — Protocol deviations | 3 | 4 | 3
Not completed — Withdrawal by Subject | 7 | 8 | 21
Not completed — Adverse Event | 16 | 18 | 23
Not completed — Abnormal test procedure | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NVA237 + Fluticasone/Salmeterol (Flu/Sal) | Tiotropium + Flu/Sal | Flu/Sal | Total
Number analyzed (Participants) | 257 | 258 | 257 | 772
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.2 (8.38) | 68.0 (7.74) | 67.8 (8.49) | 68.0 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 98 | 83 | 275
  Male | 163 | 160 | 174 | 497

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Trough Forced Expiratory Volume in 1 Second (FEV1) (NVA237 Versus Tiotropium)
Description: Spirometry was conducted according to internationally accepted standards. Trough FEV1 referred to the mean of FEV1 at 23:15 hours and 23:45 hours after the morning dose of study drug. The baseline was defined as the average of FEV1 values taken in the clinic 45 min and 15 min prior to the first dose of randomized treatment at Visit 3. A mixed model was used and contained treatment as a fixed effect with the baseline measurement of trough FEV1, FEV1 prior to inhalation of short acting bronchodilators, and FEV1 post-inhalation of bronchodilators and stratification factors as covariates. A positive change from baseline indicates improvement.
Time Frame: baseline, 12 weeks
Population: Participants from the per-protocol set (PPS), who had values at both baseline and week 12, were included in the analysis. The PPS included all randomized participants who had at least one dose of study drug and who were without any major protocol or non-protocol deviations.
Measure: Mean (Standard Error); unit: liters
Arm/Group | NVA237 + Fluticasone/Salmeterol (Flu/Sal) | Tiotropium + Flu/Sal
Number analyzed (Participants) | 194 | 185
liters | 0.095 (0.0131) | 0.102 (0.0135)

2. Secondary Outcome: Change From Baseline in Mean Trough FEV1 (Flu/Sal Versus NVA237/Tiotropium+Flu/Sal)
Description: Spirometry was conducted according to internationally accepted standards. Trough FEV1 referred to the mean of FEV1 at 23:15h and 23:45h after the morning dose of study drug. The baseline was defined as the average of FEV1 values taken in the clinic 45min and 15min prior to the first dose of randomized treatment at Visit 3. A mixed model was used and contained treatment as a fixed effect with the baseline measurement of trough FEV1, FEV1 prior to inhalation of short acting bronchodilators, and FEV1 post-inhalation of bronchodilators and stratification factors as covariates. A positive change from baseline indicates improvement.
Time Frame: baseline, 4 weeks, 8 weeks, 12 weeks
Population: Full Analysis Set: The full analysis set included all randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Error); unit: Liters
Groups:
- NVA237/Tiotropium+Flu/Sal: NVA237+Flu/Sal and Tiotropium+Flu/Sal arms
Arm/Group | Flu/Sal | NVA237/Tiotropium+Flu/Sal
Number analyzed (Participants) | 257 | 515
Liters
  Week 4 | -0.010 (0.0099) | 0.077 (0.0073)
  Week 8 | -0.002 (0.0099) | 0.088 (0.0073)
  Week 12 | -0.012 (0.0099) | 0.088 (0.0073)

3. Secondary Outcome: Change From Baseline in Mean Trough FEV1
Description: as for outcome 2
Time Frame: baseline, 4 weeks, 8 weeks, 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Liters
Arm/Group | NVA237 + Fluticasone/Salmeterol (Flu/Sal) | Tiotropium + Flu/Sal | Flu/Sal
Number analyzed (Participants) | 257 | 258 | 257
Liters
  Week 4 | 0.077 (0.0100) | 0.077 (0.0101) | -0.010 (0.0099)
  Week 8 | 0.084 (0.0100) | 0.092 (0.0101) | -0.002 (0.0099)
  Week 12 | 0.089 (0.0100) | 0.087 (0.0101) | -0.012 (0.0099)

4. Secondary Outcome: Change From Baseline in Total Score of the St George's Respiratory Questionnaire for COPD Patients (SGRQ-C) After 12 Weeks of Treatment
Description: SGRQ-C is a health related quality of life questionnaire consisting of 40 items divided into two components: 1) symptoms, 2) activity& impacts. The lowest possible value is zero and the highest is 100. Higher values corresponded to greater impairment in quality of life. An analysis model included terms for treatment, baseline total SGRQ score, FEV1 and baseline smoking status. The model also contained as fixed effects the baseline total SGRQ score, FEV1 prior to inhalation of short acting bronchodilator, FEV1 post inhalation of short acting bronchodilator and stratification factors as covariates. A negative change from baseline indicates improvement.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | NVA237 + Fluticasone/Salmeterol (Flu/Sal) | Tiotropium + Flu/Sal | Flu/Sal
Number analyzed (Participants) | 257 | 258 | 257
units on a scale | -2.806 (0.6772) | -3.902 (0.6920) | -0.652 (0.6871)

5. Secondary Outcome: Change From Baseline in the Mean Daily Number of Puffs of Rescue Medication Use
Description: The total number of puffs of rescue medication used over the last 12 h recorded in the morning (nighttime use) and in the evening (daytime use) over the full 12 weeks was divided by the total number of days with non-missing rescue data to derive the mean daytime and nighttime number of puffs of rescue medication. Change from baseline in the mean daytime and nighttime number of puffs of rescue medication was analyzed as for the change from baseline in the mean daily number of puffs of rescue medication.
Time Frame: baseline, 12 weeks
Population: Participants from the full analysis set (FAS), who had outcome measure data with applicable fixed effects/covariates according to the analysis model, were analyzed only. The full analysis set included all randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Error); unit: puffs of rescue medication
Arm/Group | NVA237 + Fluticasone/Salmeterol (Flu/Sal) | Tiotropium + Flu/Sal | Flu/Sal
Number analyzed (Participants) | 247 | 251 | 241
puffs of rescue medication | 2.191 (0.1384) | 2.093 (0.1397) | 2.908 (0.1395)

6. Secondary Outcome: Mean Percentage of Nights With 'no Nighttime Awakenings'
Description: A night with 'no nighttime awakenings' is defined from diary data as any night where patient did not wake up due to symptoms. Total number of nights with 'no nighttime awakenings' over treatment period was divided by total number of nights where diary recordings have been made in order to derive percentage of 'no nighttime awakenings' which will be summarized by treatment and analyzed using a similar mixed model as specified for primary analysis. Diary data recorded during the 7 day run-in period was used to calculate baseline percentage of nights 'no nighttime awakenings'.
Time Frame: 12 weeks
Population: as for outcome 5
Measure: Mean (Standard Error); unit: Percentage of nights
Arm/Group | NVA237 + Fluticasone/Salmeterol (Flu/Sal) | Tiotropium + Flu/Sal | Flu/Sal
Number analyzed (Participants) | 242 | 251 | 239
Percentage of nights | 0.834 (0.0124) | 0.816 (0.0124) | 0.823 (0.0124)

7. Secondary Outcome: Mean Percentage of Days With Performance of Usual Activities
Description: A 'day able to perform usual daily activities' was defined from diary data as any day where the patient was not prevented from performing their usual daily activities due to respiratory symptoms. The percentage of 'days able to perform usual daily activities' was derived and analyzed using a similar mixed model as specified for primary analysis as for the percentage of nights with 'no nighttime awakenings'.
Time Frame: 12 weeks
Population: as for outcome 5
Measure: Mean (Standard Error); unit: Percentage of days
Arm/Group | NVA237 + Fluticasone/Salmeterol (Flu/Sal) | Tiotropium + Flu/Sal | Flu/Sal
Number analyzed (Participants) | 243 | 248 | 237
Percentage of days | 0.934 (0.0087) | 0.946 (0.0088) | 0.903 (0.0088)

ADVERSE EVENTS:
Arm/Group | NVA237 + Fluticasone/Salmeterol (Flu/Sal) | Tiotropium + Flu/Sal | Flu/Sal
Serious Adverse Events (participants affected / at risk) | 15/257 | 22/258 | 15/257
Other Adverse Events (participants affected / at risk) | 114/257 | 124/258 | 111/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 + Fluticasone/Salmeterol (Flu/Sal) (N=257) | Tiotropium + Flu/Sal (N=258) | Flu/Sal (N=257)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 1
Atrial flutter (Cardiac disorders) | 1 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Breast abscess (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2 | 2
Pneumonia viral (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Femoral artery aneurysm (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 + Fluticasone/Salmeterol (Flu/Sal) (N=257) | Tiotropium + Flu/Sal (N=258) | Flu/Sal (N=257)
Palpitations (Cardiac disorders) | 0 | 3 | 0
Conjunctivitis (Eye disorders) | 0 | 3 | 3
Constipation (Gastrointestinal disorders) | 4 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 5 | 9 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3 | 2
Mouth ulceration (Gastrointestinal disorders) | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 9 | 3
Chest discomfort (General disorders) | 2 | 3 | 0
Chest pain (General disorders) | 3 | 2 | 3
Fatigue (General disorders) | 0 | 5 | 2
Oedema peripheral (General disorders) | 3 | 3 | 1
Bronchitis (Infections and infestations) | 2 | 1 | 3
Diverticulitis (Infections and infestations) | 0 | 1 | 3
Gastroenteritis (Infections and infestations) | 1 | 3 | 2
Lower respiratory tract infection (Infections and infestations) | 7 | 5 | 4
Nasopharyngitis (Infections and infestations) | 3 | 7 | 5
Oral candidiasis (Infections and infestations) | 12 | 13 | 9
Sinusitis (Infections and infestations) | 2 | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 17 | 13 | 11
Viral upper respiratory tract infection (Infections and infestations) | 3 | 4 | 5
Wound infection (Infections and infestations) | 3 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 3
Laceration (Injury, poisoning and procedural complications) | 2 | 3 | 2
Limb injury (Injury, poisoning and procedural complications) | 1 | 3 | 0
Muscle strain (Injury, poisoning and procedural complications) | 4 | 3 | 4
Weight increased (Investigations) | 3 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 8 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 9 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 2
Aphonia (Nervous system disorders) | 0 | 3 | 2
Dizziness (Nervous system disorders) | 2 | 4 | 4
Headache (Nervous system disorders) | 3 | 4 | 13
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 15 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 | 15 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 10 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 3
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Hypertension (Vascular disorders) | 3 | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.